CLINICAL TRIAL: NCT03302598
Title: Assessment of Relation Between Recurrence of Enterocutaneous Fistula and Preoperative C-reactive Protein Level After Complete Surgical Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, osama khalil, assistant professor, Zagazig University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IR-12758-2
Record Dates: First submitted 2017-09-24; First posted 2017-10-05 (Actual); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: Enterocutaneous Fistula
Keywords: enterocutaneous fistula - C-reactive protein- surgical repair
MeSH Terms: conditions — Intestinal Fistula

STUDY DESIGN:
Intervention Model Description: A prospective study of 40 patients admitted with the diagnosis of enterocutaneous fistula and prepared for definite surgical repair in the form of resection anastomosis of ECF. the investigators used preoperative serum C-reactive protein as predicting factor to recurrence and independent variable for timing of surgery.

ARMS (1):
- patients with enterocutaneous fistula (Other)
  Interventions: Diagnostic Test: serum C-reactive protein

INTERVENTIONS:
Diagnostic Test: serum C-reactive protein

SUMMARY:
A prospective study of 40 patients admitted with the diagnosis of enterocutaneous fistula and prepared for definite surgical repair in the form of resection anastomosis of ECF. The investigators used preoperative serum C-reactive protein as predicting factor to recurrence and independent variable for timing of surgery.

DETAILED DESCRIPTION:
There is a controversy in timing of operation. The timing depends on clinical assessment, laboratory tests and radiological investigations. The cornerstone of this decision is to control sepsis and inflammatory condition before surgery. This issue made surgeons favor longer interval between incidence of ECF and definite surgical treatment. In some cases there may be a hidden place for infection or continuation of the inflammatory situation without clear signs, which necessitated the presence of a possible indicator helps in making the surgical decision. Serum C-reactive protein is the common inflammatory marker used to exclude inflammatory condition. Although its level is within normal range but some cases showed high recurrence rate when the level exceeded certain as the investigators believed in their study. Now the investigators can say that the perioperative serum C-reactive protein level can be used as an objective parameter for helping to make surgical decision and reduce recurrence of ECF.

ELIGIBILITY:
Inclusion Criteria:

* patients with ECF were included in the study

Exclusion Criteria:

* Cases submitted for surgical treatment with protecting stoma or terminal were excluded from our study. Other fistulas like perianal, pancreatic, biliary and internal fistulas were not involved due to their different nature, treatment and prognosis

Ages: 56 Years to 77 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-01-20 (Actual); Primary Completion 2017-01-20 (Actual); Study Completion 2017-04-15 (Actual)

PRIMARY OUTCOMES:
C-reactive protein can be used as predicting factor for recurrence of ECF after definite surgical treatment as well as helping surgeon to take decision for proper time of operation. | 2 years
  the investigator will measure the preoperative C-reactive protein in cases of ECF which are scheduled for operative treatment . The level of c-reactive protein will be measured in the postoperative recurrent cases . we aim to find a relation between perioperative level of C-reactive protein and recurrence of ECF so it can help surgeon to choose proper time for surgical treatment to avoid recurrence of ECF

IPD SHARING:
Plan to Share IPD: Undecided